CLINICAL TRIAL: NCT00760786
Title: Effects of Intensive Lipid Lowering and Omega-3 Fatty Acid on Composition of Coronary Atherosclerotic Plaque: Serial Virtual Histology Intravascular Ultrasound Analysis
Brief Title: Effects of Intensive Lipid Lowering and Omega-3 Fatty Acid on Composition of Coronary Atherosclerotic Plaque
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Samsung Medical Center (Other)
Responsible Party: Joo-Yong Hahn, MD, PhD / Professor, Samsung Medical Center
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: SMC IRB 2007-09-006
Record Dates: First submitted 2008-09-25; First posted 2008-09-26 (Estimated); Last update posted 2008-09-26 (Estimated); Status verified 2008-09

CONDITIONS: Acute Coronary Syndrome
Keywords: IVUS-VH; Plaque characterization; Omega3-fatty acid; Atorvastatin
MeSH Terms: conditions — Acute Coronary Syndrome | interventions — Docosahexaenoic Acids

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- 1 (Active Comparator): Intensive lipid lowering plus Omega3-fatty acid
  Interventions: Drug: Intensive lipid lowering plus Omega3-fatty acid
- 2 (Active Comparator): Moderate lipid lowering plus Omega3-fatty acid
  Interventions: Drug: Moderate lipid lowering plus Omega3-fatty acid
- 3 (Active Comparator): Intensive lipid lowering plus placebo
  Interventions: Drug: Intensive lipid lowering plus placebo
- 4 (Active Comparator): Moderate lipid lowering plus placebo
  Interventions: Drug: Moderate lipid lowering plus placebo

INTERVENTIONS:
Drug: Intensive lipid lowering plus Omega3-fatty acid — Atorvastatin 40mg qd plus Omega3-fatty acid 2.0mg qd
  Arms: 1
Drug: Moderate lipid lowering plus Omega3-fatty acid — atorvastatin 10mg qd plus Omega3-fatty acid 2.0mg qd
  Arms: 2
Drug: Intensive lipid lowering plus placebo — atorvastatin 40mg qd
  Arms: 3
Drug: Moderate lipid lowering plus placebo — atorvastatin 10mg qd
  Arms: 4

SUMMARY:
The purpose of this study is to determine whether intensive lipid lowering and Omega-3 fatty acid are effective in the treatment of coronary atherosclerotic plaque.

ELIGIBILITY:
Inclusion Criteria:

* Acute coronary syndrome within 48 hours of symptom onset
* Have de novo non-culprit coronary artery stenosis 20% to 70% by visual estimation

Exclusion Criteria:

* Cardiogenic shock
* ST segment elevation myocardial infarction within 1 week
* Hematologic disorder: neutropenia (neutrophil<3000/mm3), thrombocytopenia (platelet<100,000/mm3)
* Liver enzyme elevation: serum aspartate aminotransferase or alanine aminotransferase concentrations more than 3 times the upper limit of normal
* Impaired renal function with serum creatinine > 2mg/dL
* Bleeding diathesis or history of coagulopathy
* Pregnancy
* Hypersensitivity to heparin, dye, aspirin, clopidogrel, statin, or fish

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2008-07; Primary Completion 2010-02 (Estimated)

PRIMARY OUTCOMES:
Plaque stabilization using serial virtual histology intravascular ultrasound analysis | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Joo-Yong Han, Professor, Principal Investigator — Samsung Medical Center
Locations (1):
- Cardiac and Vascular Center; Samsung Medical Center, Seoul, South Korea